CLINICAL TRIAL: NCT06189794
Title: Effects of Rosa Damascena and Frankincense Essential Oils in Labor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Tuba Kızılkaya, Asst. Prof. PhD, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20062023
Record Dates: First submitted 2023-12-16; First posted 2024-01-05 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-07

CONDITIONS: Labor Pain
Keywords: Aromatherapy; Childbirth Problems; Rosa damascena; Frankincense; Comfort
MeSH Terms: conditions — Labor Pain | interventions — Frankincense

STUDY DESIGN:
Who Masked: Participant
Masking Description: Pregnant women won't be introduced which essential oil would be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rosa damascena oil group (Experimental): Rosa Damascene oil will be used
  Interventions: Other: Rosa damascena oil
- Frankincense oil group (Active Comparator): Frankincense oil will be used
  Interventions: Other: Rosa damascena oil
- Solution group (Placebo Comparator): %0.9 NaCl Isotonical Solution will be used
  Interventions: Other: Rosa damascena oil

INTERVENTIONS:
Other: Rosa damascena oil — Essential oils will used by inhalation
  Other Names: Frankincense oil; Solution group

SUMMARY:
This randomized controlled study aims to compare effects of different essential oils in labor pain, anxiety and childbirth comfort. The main questions it aims to answer are:

Is it effective using rosa damascena oil during labor? Is it effective using frankincense oil during labor? Which essential oil is more effective during labor Researchers will compare aromatherapy oils groups to see labor pain, anxiety and childbirth comfort levels of pregnant women.

DETAILED DESCRIPTION:
During childbirth; pain, anxiety, and comfort level of women have a critical importance for a positive childbirth experience. So this study aims to compare the effects of different essential oils on labor pain, anxiety and labor comfort. In some studies, rosa damascena was found effective for labor pain. However, there are limited studies about comfort level and anxiety level of women during labor. So we aimed to investigate whether rosa damascena oil was effective for labor comfort and anxiety level or not. Samely it will be investigated frankincense oil was effective for labor comfort and anxiety level or not. Also which essential oil was more effective during labor will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant women who are at latent phase of labor

Exclusion Criteria:

* Complicated pregnancy (preeclampsia, hypertension, diabetes etc.)
* Women who will have planned cesarean section
* Asthma or any other respiratory disease
* Allergies to Rosa Damascena or Frankincense oil

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 39 (Estimated)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
labor pain | 3 hours
  Numerical Rating Score. requires the patient to rate their pain on a defined scale. 0-10 where 0 is no pain and 10 is the worst pain imaginable.
childbirth comfort | 3 hours
  Childbirth Comfort Questionnaire. It has 14 items to assess the comfort of the women during childbirth. The minimum score that can be obtained from the scale is 14 and the highest score is 70. Items 2,4,6,9,12,13,14 need to be reversed. As the score increases, high level comfort is indicated, and as it decreases, low level comfort is indicated.
anxiety | 3 hours
  Spielberger Anxiety Questionnaire. This questionnaire is a commonly used measure of trait and state anxiety. has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Kızılkaya, Asst.Prof., Principal Investigator — Balikesir University Hospital
Locations (1):
- Balikesir University Hospital, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No